CLINICAL TRIAL: NCT00678899
Title: Evaluation of the Nucleus Hybrid™ L24 Cochlear Implant
Brief Title: Evaluation of the Nucleus Hybrid™ L24 Cochlear Implant System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CORP5180
Record Dates: First submitted 2008-05-14; First posted 2008-05-16 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-06

CONDITIONS: Sensorineural Hearing Loss
Keywords: High frequency severe to profound
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgery (Experimental): Implantation with the Nucleus Hybrid L24 Cochlear Implant
  Interventions: Device: Nucleus Hybrid L24

INTERVENTIONS:
Device: Nucleus Hybrid L24 — Implantation with Nucleus Hybrid L24 cochlear implant

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy associated with the provision of acoustic and electric sound processing to individuals who demonstrate significant residual low-frequency hearing and profound high-frequency (above 1500 Hz) sensorineural hearing loss. Delivery of acoustic-electric stimulation will be provided by the Nucleus Hybrid L24 cochlear implant system.

ELIGIBILITY:
Inclusion Criteria:

1. Eighteen years of age or older at the time of implantation.
2. Severe to profound (a threshold average of 2000, 3000, & 4000 Hz > 75dB HL) sensorineural hearing loss for frequencies > 1500 Hz. Low-frequency thresholds up to and including 500 Hz should be no poorer than 60 dB HL.
3. Consonant Nucleus Consonant (CNC) monosyllabic word recognition score (mean of two lists) between 10% and 60%, inclusive (i.e., 10% <= score <= 60%), in the ear to be implanted.
4. CNC word recognition score in the contralateral ear equal to, or better than, the ear to be implanted but not more than 80%.
5. English spoken as a primary language.

Exclusion Criteria:

1. Duration of severe-to-profound hearing loss greater than 30 years.
2. Congenital hearing loss (for the purpose of this study, onset prior to 2 years-of-age).
3. Medical or psychological conditions that contraindicate undergoing surgery.
4. Ossification or any other cochlear anomaly that might prevent complete insertion of the electrode array.
5. Conductive overlay of 15 dB or greater at two or more frequencies, in the range 250 to 1000 Hz.
6. Hearing loss of neural or central origin.
7. Diagnosis of Auditory Neuropathy.
8. Active middle-ear infection.
9. Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices.
10. Unwillingness or inability of the candidate to comply with all investigational requirements.
11. Additional handicaps that would prevent or restrict participation in the audiological evaluations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-04; Primary Completion 2012-06 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John T Roland, MD, Principal Investigator — NYU MEDICAL CENTER
Locations (1):
- NYU Medical Center, New York, New York, United States

REFERENCES:
- [Derived] Reinhart PN, Parkinson AJ, Dunn CC, Gantz BJ. Factors Affecting Audiometric and Speech Perception Outcomes in Hybrid Cochlear Implant Recipients. Laryngoscope. 2025 Oct 8. doi: 10.1002/lary.70195. Online ahead of print. PMID 41059917
- [Derived] Roland JT Jr, Gantz BJ, Waltzman SB, Parkinson AJ. Long-term outcomes of cochlear implantation in patients with high-frequency hearing loss. Laryngoscope. 2018 Aug;128(8):1939-1945. doi: 10.1002/lary.27073. Epub 2018 Jan 13. PMID 29330858

RESULTS

PARTICIPANT FLOW:
Groups:
- 6 Months Post Activation: Subjects implanted with the Hybrid L implant who completed the primary endpoint of 6 months postactivation
Period: Overall Study
Arm/Group | 6 Months Post Activation
Started | 50
Completed | 49
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Surgery
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (14.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 25
Duration of hearing loss [Mean (Standard Deviation); unit: years] | 28.1 (14.9)
Duration of severe to profound high frequency hearing loss [Mean (Standard Deviation); unit: years] | 13.1 (7.2)
Monosyllabic words [Mean (Standard Deviation); unit: percent correct] — The test consists of 10 recorded lists of 50 monosyllabic words in CD format. For this study, two lists will be administered in quiet at a level equal to 60 dBA in the sound field and scored as a total number of words correct, which will be expressed as a percentage correct for this study.
  percent correct | 28.4 (14.7)
AzBio sentences [Mean (Standard Deviation); unit: percent correct] — The AzBio Sentence Test consists of 15 lists of 20 sentences each. AzBio sentences are spoken by different talkers in a conversational style with limited contextual cues that the listener can use to predict or 'fill in' unintelligible words. Each list includes 5 sentences from 4 different male and female speakers. Each word in the sentence counts towards the overall score.
  percent correct | 16.3 (14.4)

OUTCOME MEASURES:

1. Primary Outcome: Consonant Nucleus Consonant (CNC) Monosyllabic Word Score-Treated Ear (CO-PRIMARY)
Description: The co-primary study endpoints will be statistically significant differences between the mean, preoperative monosyllabic CNC word score (unilateral acoustic, ear to be implanted) and the postoperative monosyllabic CNC word scores (Hybrid mode) for the activated, Hybrid L24 cochlear implant subjects.
  The CNC Words test consists of 10 recorded lists of 50 monosyllabic words in CD format. For this study, two lists will be administered in quiet at a level equal to 60 dBA in the sound field and scored as a total number of words correct, which will be expressed as a percentage correct for this study.
Time Frame: 6 Months Postactivation
Measure: Mean (Standard Deviation); unit: percentage of words correct
Groups:
- 6 Months Postactivation: Subjects implanted with the Hybrid L implant who completed the primary endpoint of 6 months postactivation
Arm/Group | 6 Months Postactivation
Number analyzed (Participants) | 49
percentage of words correct | 65.4 (25.4)

2. Primary Outcome: AzBio Sentence Score in Noise - Treated Ear (Co-Primary)
Description: The co-primary study endpoints will be statistically significant differences between the mean, preoperative AzBio Sentences score in noise (unilateral acoustic, ear to be implanted) and postoperative AzBio Sentences score in noise (Hybrid mode) for the activated, Hybrid L24 cochlear implant subjects.
  The AzBio Sentence Test consists of 15 lists of 20 sentences each. AzBio sentences are spoken by different talkers in a conversational style with limited contextual cues that the listener can use to predict or 'fill in' unintelligible words. Each list includes 5 sentences from 4 different male and female speakers. Each word in the sentence counts towards the overall score.
Time Frame: 6 Months Postactivation
Measure: Mean (Standard Deviation); unit: percentage of words correct
Arm/Group | 6 Months Post Activation
Number analyzed (Participants) | 49
percentage of words correct | 49.2 (30.8)

3. Secondary Outcome: Consonant Nucleus Consonant (CNC) Monosyllabic Words - Treated Ear
Description: Secondary efficacy endpoints using binomial comparisons (based on the postoperative Hybrid condition) are as follows:
  The CNC Words test consists of 10 recorded lists of 50 monosyllabic words in CD format. For this study, two lists will be administered in quiet at a level equal to 60 dBA in the sound field. The percentage of subjects that scored equal to or better than they did in the pre-operative unilateral acoustic-only condition will be reported.
Time Frame: 6 Months Postactivation
Measure: Number; unit: percentage of subjects
Arm/Group | 6 Months Post Activation
Number analyzed (Participants) | 49
percentage of subjects | 96

4. Secondary Outcome: AzBio Sentence Score-Treated Ear
Description: Secondary efficacy endpoints using binomial comparisons (based on the postoperative Hybrid condition) are as follows:
  The AzBio Sentence Test consists of 15 lists of 20 sentences each. AzBio sentences are spoken by different talkers in a conversational style with limited contextual cues that the listener can use to predict or 'fill in'unintelligible words. Each list includes 5 sentences from 4 different male and female speakers. Each word in the sentence counts toward the overall score. The percentage of subjects that scored equal to or better than they did in the pre-operative acoustic only condition will be reported.
Time Frame: 6 Months Postactivation
Measure: Number; unit: percentage of subjects
Arm/Group | 6 Months Post Activation
Number analyzed (Participants) | 49
percentage of subjects | 89.9

ADVERSE EVENTS:
Arm/Group | Surgery
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 34/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery (N=50)
hearing loss (Ear and labyrinth disorders) | 22 (22)
Open/short circuited electrodes (Ear and labyrinth disorders) | 11 (11)
Increased Tinnitus (Ear and labyrinth disorders) | 6 (6)
Tinnitus not present preoperatively (Ear and labyrinth disorders) | 6 (6)
Dizziness (Ear and labyrinth disorders) | 3 (3)
Dizziness with change in hearing (Ear and labyrinth disorders) | 2 (2)
Increased tinnitus with change in hearing (Ear and labyrinth disorders) | 2 (2)
Skin irritation due to externals (Ear and labyrinth disorders) | 2 (2)
Sound quality issue (Ear and labyrinth disorders) | 2 (2)
Decrease in performance (Ear and labyrinth disorders) | 1 (1)
Imbalance (Ear and labyrinth disorders) | 1 (1)
Imbalance with change in hearing (Ear and labyrinth disorders) | 1 (1)
Increased impedances with change in hearing (Ear and labyrinth disorders) | 1 (1)
Local stitch infection (Ear and labyrinth disorders) | 1 (1)
Overstimulation (Ear and labyrinth disorders) | 1 (1)
Pain in implant ear (Ear and labyrinth disorders) | 1 (1)
Vertiginous symptoms with change in hearing (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No